CLINICAL TRIAL: NCT00647335
Title: Population Genetics of Polycystic Ovary Syndrome
Brief Title: Genetics of Polycystic Ovary Syndrome
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: University of Iowa (Other)
Responsible Party: Sponsor
Other Study IDs: 807101; University of IOWA# 200707772
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2011-11

CONDITIONS: PCOS

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Women with diagnosis of PCOS

SUMMARY:
The purpose of this study is to look at genes (DNA) and how they affect health and disease. Genes are the instruction manual for the body. The genes you get from your parents decide what you look like and how your body behaves. They can also tell us a person's risk for certain diseases and how they will respond to treatment. We will collect a saliva sample for genetic research.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is a common endocrine disorder of women, characterized by elevated levels of male hormones, absent menstruation, infrequent or very light menstruation, and reduced ability to reproduce. Genetic factors likely contribute to the etiology of PCOS, but no genes have been identified with certainty. The findings from these studies will enhance our understanding of the genetics of PCOS, a major contributor to female infertility. Better knowledge of "PCOS genes" will also help in predicting responses to treatments for infertility, insulin resistance, and other aspects of the disease.

Women with PCOS may be eligible to participate in this study if they are between the ages of 18 and 50 and have two living biological parents who are also willing to participate. Study participation involves telephone screening and consent and home collection by subjects (probands) and their parents of sputum (saliva) in a provided container. Specimen containers and signed consent forms will be returned to the study site by mail.

The major goal of this research project, the identification of genes contributing to PCOS, will provide basic understanding of the genotype-phenotype relationships that contribute to features of PCOS. Knowledge of "PCOS genes" would assist physicians in predicting and assessing responses to interventions that promote fertility, improve insulin sensitivity, and treat other aspects of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PCOS
* Both biological parents alive
* Yes to both answers and parents willing to participate

Exclusion Criteria:

* Healthy women

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women with a diagnosis of PCOS undergoing treatment at University of Pennsylvania and University of Iowa.
Sampling Method: Non-Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2008-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
PCOS gene identification. | December 2010

CONTACTS AND LOCATIONS:
Overall Officials: Anuja Dokras-Jagasia, MD, PhD, Principal Investigator — University of Pennsylvania; Brad V Voorhis, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States